CLINICAL TRIAL: NCT05842317
Title: A Randomized, Controlled, Single-center Clinical Study of Lenvatinib in Combination With Tislelizumab With or Without TACE in First-line Treatment of Advanced Hepatocellular Carcinoma.
Brief Title: Lenvatinib Plus Tislelizumab With or Without TACE in First-line Treatment of Unresectable HCC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-HCC-001
Record Dates: First submitted 2023-03-01; First posted 2023-05-06 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Lenvatinib; Tislelizumab; Transcatheter arterial chemoembolization; Efficacy; Safety
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Levatinib plus Tislelizumab (Experimental): Native-treated aHCC Patients were administered with Levatinib plus Tislelizumab
  Interventions: Drug: Lenvatinib Plus Tislelizumab
- Levatinib plus Lenvatinib with Transarterial Chemoembolization(TACE) (Experimental): Native-treated aHCC Patients were administered with Levatinib plus Tislelizumab with Transarterial Chemoembolization(TACE)
  Interventions: Drug: Lenvatinib Plus Tislelizumab; Device: Transarterial Chemoembolization(TACE)

INTERVENTIONS:
Drug: Lenvatinib Plus Tislelizumab — Lenvatinib is 12mg/d for body weight >= 60kg, 8mg/d for body weight <60kg, once daily orally, once a day, after meals (take at the same time every day as much as possible); Tislelizumab is administered intravenously at a dose of 200mg/q3w.
Device: Transarterial Chemoembolization(TACE) — A catheter is inserted through a small incision in the groin and guided to the hepatic artery, which supplies blood to the liver;A contrast dye is injected through the catheter to help visualize the blood vessels in the liver; A mixture of chemotherapy drugs and an embolic agent (such as small beads or gel foam) is injected through the catheter and into the artery that feeds the tumor;The embolic agent helps to block the blood flow to the tumor, which starves it of oxygen and nutrients; The chemotherapy drugs are then trapped in the tumor.
  Arms: Levatinib plus Lenvatinib with Transarterial Chemoembolization(TACE)

SUMMARY:
To explore the effects of lenvatinib in combination with tislelizumab with or without TACE in patients with hepatocellular carcinoma on survival, disease progression, and medication safety.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the following criteria to be included:
* Participants must voluntarily agree to participate in the study and provide written informed consent, be compliant, and agree to follow-up.
* Participants must be between 18 and 80 years old, regardless of gender, at the time of signing the informed consent form.
* Participants must be diagnosed with hepatocellular carcinoma by imaging (according to AASLD criteria or the 2022 National Health Commission Guidelines for the Diagnosis and Treatment of Liver Cancer) or histological or cytological examination.
* Patients with advanced liver cancer: patients who are in BCLC stage C or B and are eligible for TACE treatment.
* Participants must not have received systemic treatment.
* There must be at least one measurable lesion (according to RECIST 1.1 criteria, the measurable lesion must have a spiral CT scan long diameter ≥10 mm or an enlarged lymph node short diameter ≥15 mm).
* ECOG performance status must be 0-1 point within 1 week before enrollment.
* Child-Pugh liver function grade: Class A (5-6 points).
* Expected survival time ≥3 months.
* Active hepatitis B or C patients must receive relevant antiviral treatment, with HBV-DNA <2500 IU/mL (<105 copies/mL) and have received antiviral treatment for at least 14 days before participating in the study. HCV RNA-positive patients must be treated according to local standard treatment guidelines and have liver function increased no more than Grade 1 in CTCAE during treatment.
* Hematological and organ function must be adequate, based on laboratory test results obtained within 14 days before starting the study treatment, unless otherwise specified:

Complete blood count: (not transfused, not treated with G-CSF or drugs for correction) white blood cell count ≥ 3.0 x 109/L, Hb ≥ 90 g/L, neutrophil count ≥ 1.5 × 109/L, and platelet count ≥ 60 × 109/L.

* Biochemical tests: (not given albumin in the last 14 days)
* Appropriate liver function: ALB ≥ 29 g/L, ALP, ALT, and AST <5 × ULN, TBIL ≤ 3 × ULN, and PT prolongation time no more than 6s of ULN
* Appropriate renal function: Creatinine ≤ 1.5 × ULN, or creatinine clearance (CCr) >50 mL/min (using the Cockcroft-Gault formula):

Female: CrCl = ((140 - age) × body weight (kg) × 0.85) / 72 × serum creatinine (mg/dL) Male: CrCl = ((140 - age) × body weight (kg) × 1.00) / 72 × serum creatinine (mg/dL)

• Women of childbearing potential: must agree to abstain from sexual activity or use a contraceptive method with a failure rate of less than 1% for at least 6 months during the treatment period and after the last dose.

If a female patient has menstruated and has not yet reached postmenopausal status (no menstrual periods for ≥12 months continuously, and no other causes for menopause except surgical sterilization), and has not undergone sterilization surgery (removal of the ovaries and/or uterus), she is considered to be of childbearing potential.

Exclusion Criteria:

* Patients with hepatocellular carcinoma who have one or more of the following:
* Suitable for surgical treatment;
* Already underwent radical surgery with no assessable lesions;
* A history of liver transplantation or are preparing for liver transplantation.
* ECOG score ≥ 2 points.
* History of hepatic encephalopathy.
* Patients who have received systemic treatment in the past.
* Histological types of cholangiocarcinoma, sarcomatoid hepatocellular carcinoma, mixed cell carcinoma, and squamous cell carcinoma.
* Pregnant (positive pregnancy test before medication) or lactating women. Known allergy or intolerance to recombinant humanized PD-1 monoclonal antibody drugs or lenvatinib and its components (or any excipient).
* Received local anti-tumor treatment within 4 weeks before the first study drug treatment, including but not limited to surgery, radiotherapy, hepatic artery embolization, TACE, hepatic artery infusion, radiofrequency ablation, cryoablation, or percutaneous ethanol injection (palliative radiotherapy for bone metastases at least 2 weeks before study drug treatment is allowed);
* Past or current grade 3 or above digestive fistula or non-digestive fistula (such as skin) according to the CTCAE 5.0 standard.
* Various factors affecting oral administration of lenvatinib, such as inability to swallow, chronic diarrhea and intestinal obstruction, or other conditions that significantly affect drug intake and absorption.
* Clinically significant ascites (i.e., Child-Pugh score for ascites>2) or malignant ascites that require therapeutic abdominal paracentesis or drainage; or uncontrolled malignant ascites (as determined by the investigator) that cannot be controlled by diuretics or puncture.
* Major surgery (except biopsy) performed within 4 weeks before the first study drug treatment or surgical incision that has not completely healed; minor surgery (such as simple excision, biopsy, etc.) within 7 days before the first study intervention.
* Clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina pectoris, cerebrovascular accident or transient ischemic attack, congestive heart failure (New York Heart Association classification ≥2, see Appendix 4); arrhythmia requiring antiarrhythmic drugs (other than beta blockers or digoxin) for treatment; repeat electrocardiogram showing QTcF interval > 480 milliseconds (ms).
* Hepatic or renal dysfunction, such as jaundice, ascites, and/or bilirubin > 3 × ULN, creatinine ratio > 3.5 g/24 hours, or renal failure requiring blood or peritoneal dialysis. Urinalysis showing urinary protein ≥++ or confirmed 24-hour urinary protein quantification> 1.0g.
* Persistent infection of grade >2 (CTC-AE 5.0) in the past 6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | baseline up to approximately 6 months
  The proportion of patients in a clinical trial who experience either a complete response (CR), a partial response (PR) as a result of treatment.

SECONDARY OUTCOMES:
Disease control rate(DCR) | baseline up to approximately 6 months
  The proportion of patients in a clinical trial who experience either a complete response (CR), a partial response (PR), or stable disease (SD) as a result of treatment.
Progression free survival (PFS) | baseline up to approximately 12 months
  The length of time that a patient survives without their disease progressing.
Overall response (OS) | baseline up to approximately 12 months
  The length of time that a patient survives from the start of treatment until death from any cause.
Duration of Overall Response (DOR) | baseline up to approximately 6 months
  The length of time that a patient experiences a complete or partial response to treatment.
3-month/6-month PFS rate | At the time of 3-month/6-month
  The proportion of patients who survive without their disease progressing for at least 3/6 months after the start of treatment.
6-month/12-month OS rate | At the time of 6-month/12-month
  The proportion of patients who survive for at least 6/12 months after the start of treatment.
Conversion surgery rate | baseline up to approximately 12 months
  The proportion of the patients who recieved the conversion surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Nan Zhang, Beijing, Beijing Municipality, China